CLINICAL TRIAL: NCT05954026
Title: Oventus ExVent Accessory to the O2Vent Optima Device
Brief Title: Use of the ExVent Accessory With the O2Vent Optima Oral Appliance for the Treatment of Obstructive Sleep Apnea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Sleep and Chronobiology, Canada (Other)
Responsible Party: Principal Investigator, Sat Sharma, Investigator, Centre for Sleep and Chronobiology, Canada
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OVEN-02
Record Dates: First submitted 2023-07-12; First posted 2023-07-20 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Sleep Apnea, Obstructive; Sleep-Disordered Breathing
Keywords: Sleep apnea; MAD; positive expiratory pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: Prospective, open label, single-arm multicenter study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Other): Prospective, open label, single-arm multicenter study
  Interventions: Device: ExVent

INTERVENTIONS:
Device: ExVent — ExVent Accessory (inserted into the O2Vent Optima device) for treatment of sleep apnea

SUMMARY:
The ExVent is an optional accessory to the O2Vent Optima MAD and provides oral Expiratory Positive Airway Pressure (EPAP). Oral EPAP with the ExVent is designed to provide upper airway support via similar mechanisms of action of nasal EPAP devices in commercial distribution, e.g., passive dilatation of the airway, which reduces flow limitation. Nasal EPAP devices are in commercial distribution as stand-alone therapies for the treatment of OSA. The oral EPAP provided by the ExVent accessory is designed to augment the OSA therapy provided by the O2Vent Optima.

DETAILED DESCRIPTION:
Title Use of the ExVent Accessory with the O2Vent Optima Oral Appliance for the Treatment of Obstructive Sleep Apnea

Investigational Device Oventus Medical ExVent Accessory (inserted into the O2Vent Optima device)

Investigator Study Sites Up to 3 investigational sites

Regulatory Status This is a non-significant risk investigational device exemption (IDE) clinical trial. FDA approval is not required, but IRB review and approval are required.

Study Design Prospective, open label, single-arm multicenter study Sample Size Up to thirty (30) subjects will be enrolled to yield a minimum of 20 evaluable subjects (mITT subjects).

Study Objective To demonstrate that the ExVent Accessory (inserted into the O2Vent Optima device) is safe and effective in treating mild to moderate OSA Patient Population Patients who have been diagnosed with mild to moderate OSA (i.e., AHI ≥ 5 and ≤ 30)

Study Overview Study Design/ Duration:

This is a prospective, open-label, single-arm study conducted at up to 3 sites. Site participation is expected to be approximately 6 months from first subject enrollment until completion of the last study visit.

Screening Phase

1. Confirm subject meets all inclusion and exclusion criteria
2. In the absence of a prior diagnostic PSG study within the last 6 months at the investigational site's sleep lab, subject will complete a PSG study to obtain the baseline AHI and confirm a diagnosis of mild to moderate OSA

Home Use Phase

1. Subject uses the O2Vent Optima + ExVent for up to 3 months and logs usage hours.

PSG Night Subjects who successfully complete* the Home Use Phase will have an in-lab PSG sleep night while using the O2Vent Optima + ExVent

Primary Effectiveness Outcome Measure Change in AHI between baseline AHI and the AHI measured during the in-lab PSG sleep night using the O2Vent Optima + ExVent.

Primary Effectiveness Endpoint Statistically significant change in AHI with use of the O2Vent Optima + ExVent compared to baseline AHI value (i.e., no treatment).

Safety Outcome Measure Adverse events will be summarized descriptively in terms of type and frequency

Statistical Analysis This clinical trial is designed to determine whether the concomitant use of the O2Vent + ExVent devices results in a statistically significant reduction in AHI from the baseline value for each subject. A paired t-test will be used for this comparison.

A sample size calculation is based on data from a comparable group of patients (Lai, 2019), where it was determined that the mean change in AHI from baseline was -8.37, with a standard deviation of the paired differences of 7.73.

Setting alpha=0.05 and power=0.80, the calculated sample size is 9 subjects. Because of the imperfect predictability of historical data, to ensure adequate power this study will enroll 20 evaluable patients.

The mITT population will be used for this analysis**

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject aged 22 years or older.
2. Subject completed a PSG study within the last 6 months at the investigational site's sleep lab and obtained a baseline AHI confirming a diagnosis of mild to moderate obstructive sleep apnea.
3. Subject (self-reports) that he/she is currently a compliant O2Vent Optima user (i.e., using the device for at least 4 hours/night for at least 5 nights/week).
4. Subject completed initial fitting optimization of the O2Vent Optima device.
5. Investigator has determined that the subject could abstain from use of the oral appliance or other sleep apnea therapies for up to 7 days.
6. Must be able to comply with all study requirements as outlined in the protocol.

Exclusion Criteria:

Inclusion Criteria:

1. Male or female subject aged 22 years or older.
2. Subject completed a PSG study within the last 6 months at the investigational site's sleep lab and obtained a baseline AHI confirming a diagnosis of mild to moderate obstructive sleep apnea.
3. Subject (self-reports) that he/she is currently a compliant O2Vent Optima user (i.e., using the device for at least 4 hours/night for at least 5 nights/week).
4. Subject completed initial fitting optimization of the O2Vent Optima device.
5. Investigator has determined that the subject could abstain from use of the oral appliance or other sleep apnea therapies for up to 7 days.
6. Must be able to comply with all study requirements as outlined in the protocol.

Exclusion Criteria:

1. Oral cavity infection or any other oral or dental condition or problem that would limit patient use of the O2Vent Optima oral appliance.
2. Any concomitant diagnosed or suspected sleep disorder including insomnia or central apnea.
3. History of any prior OSA surgical treatments including RF ablation treatment or palatal stent devices.
4. Concomitant use of any other prescription device for treatment of OSA.
5. Female of child-bearing age who is pregnant or intending to become pregnant during the study participation period.
6. Subject with significant change in weight since completion of the diagnostic baseline PSG study (i.e., ±10% or greater change in total body weight.
7. Subject on a non-stable dose of medications or other agents that may affect sleep and/or PSG (e.g., sedatives or hypnotics).
8. Subject who consumes > 500 mg caffeine per day (e.g., > 8 cola-type beverages, > 5 cups of coffee).
9. Subject who consumes > 3 alcoholic drinks/day.
10. Subject currently enrolled in any other research study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2024-12-08 (Estimated); Study Completion 2025-03-10 (Estimated)

PRIMARY OUTCOMES:
Change in AHI between baseline AHI and the AHI measured during the in-lab PSG sleep night using the O2Vent Optima + ExVent. | Two Years
  To demonstrate that the ExVent Accessory (inserted into the O2Vent Optima device) is safe and effective in treating mild to moderate OSA. Statistically significant change in AHI with use of the O2Vent Optima + ExVent compared to baseline AHI value (i.e., no treatment).

SECONDARY OUTCOMES:
Adverse events will be summarized descriptively in terms of type and frequency | Two years
  Adverse events which might occur or have been known to occur with Mandibular Advancement devices include but are not limited to the following:
  * Tooth movement, discomfort, pain or changes in dental occlusion
  * Loss of dental restorations
  * Dental soreness
  * Pain or soreness to the temporomandibular joint
  * Excessive salivation
  * Cheek or tongue pain
  * Jaw discomfort, pain or jaw set
  * Gingivitis
  * Dry mouth
  * Difficulty sleeping

CONTACTS AND LOCATIONS:
Overall Officials: Sat Sharma, Principal Investigator — Centre for Sleep
Locations (1):
- Centre for Sleep and Chronobiology, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No